CLINICAL TRIAL: NCT04427384
Title: A Multicenter Observational Study of GammaTile™ Surgically Targeted Radiation Therapy (STaRT) in Intracranial Brain Neoplasms
Brief Title: Registry of Patients With Brain Tumors Treated With STaRT (GammaTiles)
Status: Recruiting | Type: Observational
Sponsor: GT Medical Technologies, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: GTM-101
Record Dates: First submitted 2020-06-05; First posted 2020-06-11 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Brain Tumor, Recurrent; Brain Tumor; Brain Tumor, Primary; Brain Tumor - Metastatic; Brain Tumor, Adult: Glioblastoma; Brain Tumor, Adult Meningioma
MeSH Terms: conditions — Brain Neoplasms; Meningioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- GammaTile: Patients who have received permanent implants of GammaTile radiation therapy immediately following brain tumor resection.
  Interventions: Device: GammaTile

INTERVENTIONS:
Device: GammaTile — Surgically Targeted Radiation Therapy

SUMMARY:
The objectives of this registry study are to evaluate real-world clinical outcomes and patient reported outcomes that measure the effectiveness and safety of STaRT.

DETAILED DESCRIPTION:
Patients (N=600) with surgically resected (R) brain tumors of any pathology who have undergone STaRT are eligible. Data collected will include local control, overall survival, QOL, neurocognition, functional decline, and surgical and radiation associated AE's. Data will be collected at 1, 3, 6, 9,12, 18 and 24 months, then every 6 months through 5 years. RESULT: Data will be used to benchmark clinical outcomes of STaRT therapy and allow for comparisons to existing standard-of-care treatments. This will be the first observational registry study of R+STaRT, delivered by Cs-131 sources in permanently implanted resorbable collagen tile carriers. The outcome measures captured will allow for evaluation of the potential risks and benefits of this treatment approach for patients in a real-world setting.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who undergo maximum safe resection of intracranial neoplasm(s) AND implantation of GammaTiles.
2. Willing and able to provide informed consent and to participate in all evaluations.

Exclusion Criteria:

1. Inability to undergo pre-operative and post-operative imaging for disease and implant assessment.
2. Major medical or psychiatric illness, which, in the investigator's opinion would prevent completion of treatment, ability to complete assessments at the time of enrollment, and/or interfere with follow ups.
3. Subjects who, in the investigator's opinion, are unable to understand the protocol or to give informed consent, have a history of poor cooperation, noncompliance with medical treatment, or difficulty in returning for follow up care. A legally authorized representative may provide consent if the potential subject lacks the capacity to provide consent themselves.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who received STaRT (GammaTile) intraoperatively.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2020-09-11 (Actual); Primary Completion 2028-10-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Surgical Bed-Recurrence Free Survival in Metastatic Tumor Subjects | 12 months
  No contrast enhancement in the area of the surgical bed
Surgical Bed-Recurrence Free Survival in Meningioma Tumor Subjects | 3 years
  No contrast enhancement in the area of the surgical bed
Overall Survival in High Grade Glioma Subjects | 9 months
  Median duration of survival of subjects following surgical resection of tumor

CONTACTS AND LOCATIONS:
Overall Officials: Michael A. Garcia, MD, MS, Study Director — GT Medical Technologies
Locations (53):
- United States (53):
  - HonorHeath Scottsdale Osborn Medical Center, Phoenix, Arizona
  - University of Arkansas Medical Center, Little Rock, Arkansas
  - Eden Medical Center, Castro Valley, California
  - UCSD Moores Cancer Center, La Jolla, California
  - MemorialCare Health System, Laguna Hills, California
  - Desert Regional Medical Center, Palm Springs, California
  - California Pacific Medical Center, Sutter health, San Francisco, California
  - Centura, Denver, Colorado
  - Colorado Brain & Spine Institute: Swedish Campus, Englewood, Colorado
  - BayCare Health, Clearwater, Florida
  - Ascension St. Vincent's, Jacksonville, Florida
  - Miami Cancer Institute, Baptist Health South Florida, Miami, Florida
  - Advent Health Orlando, Orlando, Florida
  - Orlando Health, Orlando, Florida
  - Florida Health Sciences Center, Inc. d/b/a Tampa General Hospital, Tampa, Florida
  - Cleveland Clinic Florida- Weston, Weston, Florida
  - Piedmont Healthcare, Atlanta, Georgia
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - St. Alphonsus Regional Medical Center, Boise, Idaho
  - Goodman Campbell Brain and Spine, Carmel, Indiana
  - Indiana University, IU Health Methodist Hospital, Indianapolis, Indiana
  - KUMC Dept of Neurosurgery, Kansas City, Kansas
  - Univeristy of Louisville Health, Louisville, Kentucky
  - Norton Cancer Institute, Louisville, Kentucky
  - Willis-Knighton Medical Center, Shreveport, Louisiana
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - University of Nebraska, Omaha, Nebraska
  - Clinical Research dep. Davison Place. Englewood Health, Englewood, New Jersey
  - Albany Medical Center, Albany, New York
  - Mount Sinai Hospital, New York, New York
  - SUNY Upstate Medical Center, Syracuse, New York
  - Montefiore Einstein, The Bronx, New York
  - Westchester Medical Center, Valhalla, New York
  - University of North Carolina Health, Chapel Hill, North Carolina
  - Vidant Heath - ECU Medical Center, Greenville, North Carolina
  - Atlantic Brain & Spine, Wilmington, North Carolina
  - Mayfield Brain and Spine, Cincinnati, Ohio
  - Kettering Health, Kettering, Ohio
  - St Luke's University Health, Sacred Heart Campus, Allentown, Pennsylvania
  - Penn State Health, Hershey, Pennsylvania
  - Allegheny Health Network, Pittsburgh, Pennsylvania
  - Brown University Health, Providence, Rhode Island
  - CHI Memorial Hospital, CommonSpirit, Chattanooga, Tennessee
  - UT Southwestern Simmons Cancer Center, Dallas, Texas
  - Baylor St. Luke's Medical Center | Baylor College of Medicine, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - University of Texas Health Science Center of San Antonio, San Antonio, Texas
  - Texas Oncology-The Woodlands, The Woodlands, Texas
  - INOVA Health, Fairfax, Virginia
  - Virginia Mason, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No